CLINICAL TRIAL: NCT02599896
Title: VRC 606: A Phase 1, Dose-Escalation Study of the Safety and Pharmacokinetics of a Human Monoclonal Antibody, VRC-HIVMAB080-00-AB (VRC01LS) and VRC-HIVMAB060-00-AB (VRC01), Administered Intravenously or Subcutaneously to Healthy Adults
Brief Title: Safety and Pharmacokinetics of a Human Monoclonal Antibody, VRC-HIVMAB080-00-AB (VRC01LS), With Broad HIV-1 Neutralizing Activity, Administered Intravenously or Subcutaneously to Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 160018; 16-I-0018
Record Dates: First submitted 2015-11-06; First posted 2015-11-09 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2018-07-25

CONDITIONS: Prevention of HIV Infection; HIV Antibodies; Monoclonal Antibody, Human; Neutralizing Antibody
Keywords: Dose Escalation; HIV Prevention; Broadly HIV-1 Neutralizing Activity; Open-Label; Half-Life
MeSH Terms: interventions — VRC01 monoclonal antibody

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes

ARMS (8):
- Group 1 (Experimental): 5 mg/kg/IV on Day 0
  Interventions: Biological: VRC-HIVMAB080-00-AB (VRC01LS)
- Group 2 (Experimental): 5 mg/kg SC on Day 0
  Interventions: Biological: VRC-HIVMAB080-00-AB (VRC01LS)
- Group 3 (Experimental): 20 mg/kg IV on Day 0
  Interventions: Biological: VRC-HIVMAB080-00-AB (VRC01LS)
- Group 4 (Experimental): 40 mg/kg IV on Day 0
  Interventions: Biological: VRC-HIVMAB080-00-AB (VRC01LS)
- Group 5 (Experimental): 5 mg/kg SC on Day 0, Week 12 and Week 24
  Interventions: Biological: VRC-HIVMAB080-00-AB (VRC01LS)
- Group 6 (Experimental): 20 mg/kg IV on Day 0, Week 12 and Week 24
  Interventions: Biological: VRC-HIVMAB080-00-AB (VRC01LS)
- Group 7 (Experimental): 5 mg/kg SC on Day 0, Week 4
  Interventions: Biological: VRC-HIVMAB060-00-AB (VRC01)
- Group 8 (Experimental): 20 mg/kg IV on Day 0, Week 4
  Interventions: Biological: VRC-HIVMAB060-00-AB (VRC01)

INTERVENTIONS:
Biological: VRC-HIVMAB080-00-AB (VRC01LS) — VRC01LS is an Investigational Monoclonal Antibody targeted to the CD4 binding site of HIV-1.
  Arms: Group 1; Group 2; Group 3; Group 4; Group 5; Group 6
Biological: VRC-HIVMAB060-00-AB (VRC01) — VRC01 is an Investigational Monoclonal Antibody targeted to the CD4 binding site of HIV-1.
  Arms: Group 7; Group 8

SUMMARY:
Background:

Antibodies help the body fight infection. VRC01LS is an antibody directed against HIV virus. HIV attacks the immune system. In animals, VRC01LS inactivated many types of HIV viruses. Researchers want to see if it does this in people.

Objectives:

To see if VRC01LS is safe and well-tolerated in people. To see what level of VRC01LS is maintained in people and if they develop an immune response to it.

Eligibility:

Healthy people ages 18 to 50

Design:

Participants will be screened in protocol number VRC 500 (NIH 11-I-0164) with medical history, physical exam, and blood and urine tests.

The study will last 24 to 48 weeks. Visits will last 2 to 8 hours.

Participants will get VRC01LS through either:

* A needle in an arm vein or
* A small needle placed into the fatty tissue under the skin of the abdomen, thigh, or arm.

Participants will be assigned to 1 of 6 groups.

Groups 1 to 4 will get 1 dose of VRC01LS. They will have follow-up visits through week 24.

Groups 5 and 6 will get 1 dose of VRC01LS every 12 weeks (3 doses). They will have 4 to 5 visits between the second and third dose, and follow-up visits through week 48.

Participants will have 1 to 3 follow-up visits in the week after receiving VRC01LS. They will record their temperature and keep a diary of symptoms for 3 days after a dose. They may have additional unscheduled visits.

At each visit, participants will have a physical exam and may have blood and urine tests.

DETAILED DESCRIPTION:
VRC 606: A Phase 1, Dose-Escalation Study of the Safety and Pharmacokinetics of a Human Monoclonal Antibody, VRC-HIVMAB080-00-AB (VRC01LS), and VRC-HIVMAB060-00-AB (VRC01), Administered Intravenously or Subcutaneously to Healthy Adults.

Study Design: This is the first study of the VRC-HIVMAB080-00-AB (VRC01LS) monoclonal antibody (MAb) in healthy adults. It is a dose-escalation study to examine safety, tolerability, dose, and pharmacokinetics of VRC01LS. The hypothesis is that VRC01LS will be safe to administer to healthy adults by the intravenous (IV) and subcutaneous (SC) routes. The secondary hypothesis is that VRC01LS will be detectable in human sera with a definable half-life. With protocol amendment, Group 7 and Group 8 were added to the protocol Version 2.0 to evaluate VRC01 and VRC01LS safety and pharmacokinetics in the same study.

Product Description: VRC-HIVMAB080-00-AB (VRC01LS) and VRC-HIVMAB060-00-AB (VRC01) are human MAb targeted to the CD4 binding site of HIV-1. VRC01LS is a modification of the VRC01 MAb (which has been shown to be safe in human studies) with the addition of the LS , 2-amino acid mutation designed to improve the half-life of the antibody. VRC01LS and VRC01 were developed by VRC/NIAID/NIH and manufactured under cGMP at the VRC Pilot Plan operated under contract by the Vaccine Clinical Material Program operated for NIAID/VRC by Leidos Biomedical Research, Inc., Frederick, MD. Vials are provided at 100 mg/mL.

Subjects: Healthy adults, 18-50 years of age.

Study Plan: There are 4 open-label, dose escalation groups (Groups 1-4) to assess VRC01LS administered IV and SC once per subject. 2 open-label groups (Groups 5 and 6) to assess VRC01LS at 5 mg/kg SC or at 20 mg/kg IV administered every 12 weeks for a total of 3 administrations per subject, and 2 open-label groups (Groups 7 and 8) to assess VRC01 at 5 mg/kg SC or at 20 mg/kg IV administered every 4 weeks for a total of 2 administrations per subject. Subjects will be randomized into Group 1 or Group 2 at a 1:1 ratio, or directly enrolled into Groups 3-6 per the dose escalation and safety evaluation plan. Enrollments into Group 7 and Group 8 will be randomized at a 1:1 ratio.

Study Duration: Subjects will be followed for 24 weeks after the last study product administration.

ELIGIBILITY:
* INCLUSION CRITERIA:

A volunteer must meet all of the following criteria:

1. Able and willing to complete the informed consent process.
2. 18 to 50 years of age.
3. Based on history and examination, must be in general good health without history of any of the conditions listed in the exclusion criteria.
4. Willing to have blood samples collected, stored indefinitely, and used for research purposes.
5. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.
6. Screening laboratory values within 84 days prior to enrollment must meet the following criteria:

   * WBC 2,500-12,000/mm(3).
   * WBC differential either within institutional normal range or accompanied by the Principal Investigator (PI) or designee approval.
   * Platelets = 125,000 to 400,000/mm(3).
   * Hemoglobin within institutional normal range.
   * Creatinine less than or equal to 1.1 x ULN.
   * ALT less than or equal to 1.25 x ULN.
   * Negative for HIV infection by the FDA approved method of detection.

   Female-Specific Criteria:
7. If a woman is secually active with a male partner and has no history of hysterectomy, tubal ligation, or menopause, then she agrees to use either a prescription birth control method or barrier birth control method from the time of study enrollment until the last study visit, or to have a monogamous partner who has had a vasectomy.
8. Negative beta-HCG (human chorionic gonadotropin) pregnancy test (urine or serum) on day of enrollment for women presumed to be of reproductive potential.

EXCLUSION CRITERIA:

A volunteer will be excluded if one or more of the following conditions apply:

1. Previous receipt of monoclonal antibody whether licensed or investigational.
2. Weight >115 kg.
3. History of a severe allergic reaction with generalized urticaria, angioedema or anaphylaxis within the 2 years prior to enrollment that has a reasonable risk of recurrence.
4. Hypertension that is not well controlled.
5. Woman who is breast-feeding, or planning to become pregnant during the study participation.
6. Receipt of any investigational study agent within 28 days prior to enrollment.
7. Any other chronic or clinically significant medical condition that in the opinion of investigator would jeopardize the safety or rights of the volunteer. Including, but not limited to: diabetes mellitus type I, chronic hepatitis; OR clinically significant forms of: drug or alcohol abuse, asthma, autoimmune disease, psychiatric disorders, heart disease, or cancer.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2015-11-16; Primary Completion 2018-07-25 (Actual); Study Completion 2018-07-25 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of VRC-HIVMAB080-00-AB administered as a single dose at 5 mg/kg IV,20 mg/kg IV,40 mg/kg IV, and 5 mg/kg SC to healthy adults | Through 24 weeks of study participation.
Evaluate the safety and tolerability of VRC-HIVMAB080-00-AB administered at 20 mg/kg IV by repeat dosing every 12 weeks for a total of 3 infusions to healthy adults. | Through 48 weeks of study participation.
Evaluate the safety and tolerability of VRC-HIVMAB080-00-AB administered at 5 mg/kg SC by repeat dosing every 12 weeks for a total of 3 injections to healthy adults. | Through 48 weeks of study participation.

SECONDARY OUTCOMES:
To evaluate the pharmacokinetics of VRC-HIVMAB080-00-AB at each dose level. | Through 24 weeks after the last dose.
To determine whether anti-drug antibody (ADA) to VRC01LS can bedetected in recipients of VRC-HIVMAB080-00-AB. | Through 24 weeks after the last dose.

CONTACTS AND LOCATIONS:
Overall Officials: Martin R Gaudinski, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Wu X, Yang ZY, Li Y, Hogerkorp CM, Schief WR, Seaman MS, Zhou T, Schmidt SD, Wu L, Xu L, Longo NS, McKee K, O'Dell S, Louder MK, Wycuff DL, Feng Y, Nason M, Doria-Rose N, Connors M, Kwong PD, Roederer M, Wyatt RT, Nabel GJ, Mascola JR. Rational design of envelope identifies broadly neutralizing human monoclonal antibodies to HIV-1. Science. 2010 Aug 13;329(5993):856-61. doi: 10.1126/science.1187659. Epub 2010 Jul 8. PMID 20616233
- [Background] Rudicell RS, Kwon YD, Ko SY, Pegu A, Louder MK, Georgiev IS, Wu X, Zhu J, Boyington JC, Chen X, Shi W, Yang ZY, Doria-Rose NA, McKee K, O'Dell S, Schmidt SD, Chuang GY, Druz A, Soto C, Yang Y, Zhang B, Zhou T, Todd JP, Lloyd KE, Eudailey J, Roberts KE, Donald BR, Bailer RT, Ledgerwood J; NISC Comparative Sequencing Program; Mullikin JC, Shapiro L, Koup RA, Graham BS, Nason MC, Connors M, Haynes BF, Rao SS, Roederer M, Kwong PD, Mascola JR, Nabel GJ. Enhanced potency of a broadly neutralizing HIV-1 antibody in vitro improves protection against lentiviral infection in vivo. J Virol. 2014 Nov;88(21):12669-82. doi: 10.1128/JVI.02213-14. Epub 2014 Aug 20. PMID 25142607
- [Background] Ko SY, Pegu A, Rudicell RS, Yang ZY, Joyce MG, Chen X, Wang K, Bao S, Kraemer TD, Rath T, Zeng M, Schmidt SD, Todd JP, Penzak SR, Saunders KO, Nason MC, Haase AT, Rao SS, Blumberg RS, Mascola JR, Nabel GJ. Enhanced neonatal Fc receptor function improves protection against primate SHIV infection. Nature. 2014 Oct 30;514(7524):642-5. doi: 10.1038/nature13612. Epub 2014 Aug 13. PMID 25119033
- [Derived] Gaudinski MR, Coates EE, Houser KV, Chen GL, Yamshchikov G, Saunders JG, Holman LA, Gordon I, Plummer S, Hendel CS, Conan-Cibotti M, Lorenzo MG, Sitar S, Carlton K, Laurencot C, Bailer RT, Narpala S, McDermott AB, Namboodiri AM, Pandey JP, Schwartz RM, Hu Z, Koup RA, Capparelli E, Graham BS, Mascola JR, Ledgerwood JE; VRC 606 Study Team. Safety and pharmacokinetics of the Fc-modified HIV-1 human monoclonal antibody VRC01LS: A Phase 1 open-label clinical trial in healthy adults. PLoS Med. 2018 Jan 24;15(1):e1002493. doi: 10.1371/journal.pmed.1002493. eCollection 2018 Jan. PMID 29364886